CLINICAL TRIAL: NCT05567692
Title: Descendance Cohort: Follow-up of Subjects With Type 2 Diabetes or at Risk of Type 2 Diabetes Defined by the Existence of the Disease in the Family in Two Successive Generations
Brief Title: Subjects With T2D or at Risk of T2D Cohort Follow-up
Acronym: DESCENDANCE
Status: Active, not recruiting | Type: Observational
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Collaborators: Institut Pasteur de Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01538-35
Record Dates: First submitted 2022-09-22; First posted 2022-10-05 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes ; Risk Prediction ; Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T2D group: subjects with type 2 diabetes
  Interventions: Other: Questionnaire
- Non-T2D group: healthy subjects
  Interventions: Diagnostic Test: OGTT; Other: HbA1c; Other: Questionnaire

INTERVENTIONS:
Diagnostic Test: OGTT — Oral Glucose Tolerance Test
  Groups: Non-T2D group
Other: HbA1c — HbA1c measurement
  Groups: Non-T2D group
Other: Questionnaire — Follow-up questionnaire

SUMMARY:
The main objective of this study is to prospectively follow the subjects included in "Descendance" cohort and to describe the occurrence of type 2 diabetes in non-diabetic subjects, which will allow us to iteratively update the "Descendance" Type 2 Diabetes risk prediction model.

DETAILED DESCRIPTION:
High risk families will be prospectively follow in order to better understand the risk of transmission of type 2 diabetes from one generation to another. The cohort will also allow us to collect additional data on diabetic patients.

The monitoring of the cohort will take place for at least 10 years with a follow-up of all participants every three years. To detect individuals who develop dysglycemia during the study, a glucose tolerance test (GTT) and HbA1c measurement will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have participated in the Descendance study
* Subjets who sign informed consent to participate in the study

Exclusion Criteria:

* Subjects not enrolled in Descendance study
* Subjects refusing to participate
* Pregnant or breastfeeding
* Subjects in emergency situations, under legal protection or unable to provide informed -consent
* Subjects lost to follow-up or died

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects included in the DESCENDANCE clinical trial (Id: NCT01727349) between 20011 and 2020, will be re-invited to participate in the Descendance cohort follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 837 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2032-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Type 2 diabetes incidence in Descendance population | 9years
  Presence of type 2 diabetes mellitus, on basis of self-reported (physician diagnosis) or diagnosed by OGTT and HbA1c

SECONDARY OUTCOMES:
Provide estimates of prevalence of diabetes and prediabetes in Descendance population | at baseline, 3-, 6- and 9-years follow-up
  To estimate the prevalence of undiagnosed diabetes mellitus and pre-diabetes in Descendance population
Study of interactions between risk factors on type 2 diabetes incidence | at baseline, 3-, 6- and 9-years follow-up
  Self-administered questionnaire. "Descendance" specific questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CHARPENTIER, Dr, Principal Investigator — Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète
Locations (1):
- Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète, Évry, France

IPD SHARING:
Plan to Share IPD: No